CLINICAL TRIAL: NCT04466878
Title: Prognostic Value of Implementing VCE on Top in Constitutional VWD-patients With GI-bleeding
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020 02
Record Dates: First submitted 2020-07-06; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-02

CONDITIONS: Von Willebrand Diseases
Keywords: Gastrointestinal bleeding; Videocapsule endoscopy; Angiodysplasia
MeSH Terms: conditions — von Willebrand Diseases; Gastrointestinal Hemorrhage; Angiodysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Citrate poor-platelet plasmaPlasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inclusion criteria: Only constitutional VWD-patients fulfilling the inclusion criteria of the French reference center for VWD will be included. Patients with acquired von Willebrand syndrome will not be included.

Material and Methods: A 15-items survey that will be sent to the 30 centers involved in the French network for bleeding disorders (MHEMO) to identify VWD-patients referred for endoscopic exploration of at least one GI-bleeding from January 2015 to December 2017. Only constitutional VWD-patients fulfilling the inclusion criteria of the French reference center for VWD will be included. Constitutional VWD diagnosis will be confirmed confirmed centrally in all patients by the French reference center for von Willebrand disease. A GI-bleeding episode will be defined as any overt or occult GI-bleeding (unexplained chronic iron deficiency anemia causing a drop of hemoglobin level by more than 2 g/dL from baseline). We will analyze patient characteristics, GI-bleeding pattern, VWD type/subtype, nature (gastroscopy, colonoscopy or VCE) and results of the endoscopic exploration and management that was applied: endoscopic therapy by argon plasma coagulation, on-demand/prophylactic-VWF replacement therapy, use of antiangiogenic drugs. If angiodysplasia without another bleeding source is identified, GI-bleeding will be categorized as angiodysplasia, if another lesion is identified GI-bleeding will be categorized as "no-angiodysplasia" and if no bleeding source is identified, GI-bleeding will be categorized as obscure GI-bleeding. Recurrence will be defined as evidence of overt GI-bleeding or a drop of hemoglobin level by more than 2 g/dL from baseline.

ELIGIBILITY:
Inclusion Criteria:

- At least one overt or occult GI-bleeding (unexplained iron deficiency anemia causing a drop of hemoglobin level by more than 2g/dL from baseline) episode between January 1st 2015 and December 31th 2017

Exclusion Criteria:

* acquired Von Willebrand syndrome

Age Groups: Child, Adult, Older Adult
Study Population: - VWD-patients fulfilling the inclusion criteria of the French reference center for VWD
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnosis yield of an endoscopic strategy including video capsule on top of conventional endoscopy | 3-years follow-up
  Diagnosis yield of an endoscopic strategy including video capsule on top of conventional endoscopy compared to conventional endoscopy alone in VWD-patients with GI-bleeding

SECONDARY OUTCOMES:
Risk prediction of GI-bleeding recurrence with videocapsule endoscopy | 2-years follow-up
  Recurrence-free survival after the first GI-bleeding event according to the presence of angiodysplasia on videocapsule endoscopy